CLINICAL TRIAL: NCT06520371
Title: Comparison of Percutaneous and Conventional Radiofrequency Applications for the Treatment of Knee Osteoarthritic Pain: A Randomized Controlled Trial
Brief Title: Percutaneous vs Conventional Radiofrequency Applications for the Treatment of Knee Osteoarthritic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR670/4/24
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous; Conventional; Radiofrequency; Knee Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous radiofrequency group (Experimental): Patients will receive percutaneous radiofrequency.
  Interventions: Device: Percutaneous radiofrequency
- Conventional radiofrequency group (Active Comparator): Patients will receive conventional radiofrequency.
  Interventions: Device: Conventional radiofrequency

INTERVENTIONS:
Device: Percutaneous radiofrequency — For the percutaneous radiofrequency treatment, a medium electrode size will be placed on either side of the knee: one skin electrode on the inside and one on the outside of the knee for 15 minutes.
  Arms: Percutaneous radiofrequency group
Device: Conventional radiofrequency — For the conventional radiofrequency treatment, a 50 Hz sensory stimulation will be performed with a 10 cm, 22 gauge, 10 mm active tip radiofrequency cannula. After receiving the appropriate sensory and motor stimuli, a radiofrequency of 90°C will be applied for 90 s.
  Arms: Conventional radiofrequency group

SUMMARY:
This study aims to compare percutaneous and conventional radiofrequency applications for the treatment of knee osteoarthritic pain.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive degenerative joint disease that affects the joint cartilage and surrounding tissues. It mostly affects the weight-bearing joints, and in this respect, the knee joint is one of the joints that is most affected.

Radiofrequency (RF) treatment has been used for several painful conditions such as trigeminal neuralgia, cancer pain, and spinal pain. To destroy nerves or disrupt the transmission of pain signals, originally using producing heat lesions, RF current is applied to the trigeminal ganglion, the spinothalamic tracts of the spinal cord, the medial branches of posterior rami, and the dorsal root ganglion. In addition to these, there have been a few attempts to apply RF current for the treatment of painful conditions of joints of the extremities.

Percutaneous radiofrequency ablation (RFA) of articular sensory nerves has recently emerged as an attractive and minimally invasive approach to treat chronic pain due to large-joint osteoarthritis in select patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Both sexes.
* Patients with knee osteoarthritis.
* Previous conservative treatments longer than 3 months.
* Visual analog scale (VAS)≥ 4.
* Radiological osteoarthritis grades 3 and 4 according to the Kellgren-Lawrence grading system (0 = none, 1 = doubtful, 2 = minimal, 3 = moderate, and 4 = severe).

Exclusion Criteria:

* Prior knee surgery.
* Allergies to local anesthetics.
* Connective tissue diseases affect the knee.
* Serious neurologic or psychiatric disorders.
* Injection with steroids or hyaluronic acids during the previous 3 months.
* History of septic arthritis.
* Sciatic pain.
* Cardiac pacemaker users.
* Anticoagulant medications.
* Prior electroacupuncture treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 12th week post-procedure
  Degree of pain will be assessed using visual analog scale (VAS). Each patient will obtain a score between 0 and 10 (Zero means no pain, and ten means the worst pain). VAS will be assessed pre-procedure and post-procedure 2nd, 6th, and 12th week.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores | 12th week post-procedure
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores: range from 0 to 96 (0 represents the best health status and 96 the worst possible status). The higher the score, the poorer the function. It will be assessed pre-procedure and post-procedure 1, 4, and 12th week.
Patient satisfaction | 12th week post-procedure
  Degree of patient satisfaction will be assessed on a 5-point Likert scale Patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied ; 5, extremely satisfied). It will be assessed pre-procedure and post-procedure 1, 4, and 12th week.
Incidence of adverse events | 12th week post-procedure
  Incidence of adverse events such as bleeding, neurological damage, infection, abnormal proprioception, numbness, paresthesia, and motor weakness will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.